CLINICAL TRIAL: NCT03847766
Title: Tele Follow-up Using Patient-reported Outcomes (PRO) Measures in Patients With Chronic Kidney Disease - the PROKID Study
Brief Title: Follow-up Using Patient-Reported Outcome (PRO) Measures in Patients With Chronic Kidney Disease
Acronym: PROKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regional Hospital West Jutland (Other); Aarhus University Hospital (Other); TrygFonden, Denmark (Industry); Karen Elise Jensen Foundation (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROKID
Record Dates: First submitted 2019-01-23; First posted 2019-02-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Diseases
Keywords: PRO-based follow-up, TelePRO; Outpatients, Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The randomization will be done by the AmbuFlex-system (a generic on-line system for self-recorded patient reported outcomes) as a part of the inclusion process.
  Patients in the intervention arms will receive diagnosis specific questionnaires through a safe internet connection every third month. The responses are seen by the clinicians in the Electronic Health Record.
  Patients will receive 2 reminders if they do not answer the questionnaires and clinicians will call the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRO-based follow-up (Experimental): Patients will receive a questionnaire every 3 months. The PRO questionnaire is used as decision aid together with other available clinical data to decide whether the patient needs a visit or not. Hence, patients only visit the outpatient clinic if there is a clinical need or a patient's wish. The actual response for each questionnaire automatically results in a colour code (green, yellow or red). A red or yellow response indicates that the patient needs to be contacted. A green colour indicates no need for a visit. Based on an overview of the questionnaire and the patient's blood samples a physician decides whether this patient should have a telephone consultation or the patient needs to be seen in the clinic.
  Interventions: Behavioral: PRO-based follow-up
- PRO-based telephone consultations (Experimental): Patients receive an electronic questionnaire every 3 months prior to a scheduled telephone consultation.The PRO questionnaire is used as dialogue support during the telephone consultation. The actual response for each item automatically results in a colour code (green, yellow or red). A red response indicates that the patient has a problem; a yellow colour indicates a potential problem, while a green colour indicates no problems.
  Interventions: Behavioral: PRO-based telephone consultation
- Usual outpatient follow-up visits (No Intervention): Patients in the control group will continue to have usual scheduled outpatient follow-up visits at the hospital initiated by the physician every 3 months. These patients do not use the clinical PRO questionnaire, but complete the research questionnaires.

INTERVENTIONS:
Behavioral: PRO-based follow-up — Diagnose specific questionnaires are used to screen patients in need of contact to the outpatient clinic
  Other Names: TelePRO
  Arms: PRO-based follow-up
Behavioral: PRO-based telephone consultation — diagnose-specific questionnaires are used to support communication between clinician and patient during a phone consultation
  Arms: PRO-based telephone consultations

SUMMARY:
This randomized controlled trial (RCT) will evaluate if PRO-based follow-up is at least as effective as usual outpatient follow-up in managing decline in renal function and maintaining patients' quality of life. Furthermore, we intend to characterize the target patient group that is suitable for PRO-based follow up in a group of patients suffering from renal insufficiency.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the use of Patient-reported Outcome (PRO) follow-up among patients with chronic kidney disease. Usual outpatient follow-up visits will be replaced with diagnosis-specific electronic questionnaires filled in by the patient at home. Participants in the PRO-based follow up will complete a disease specific questionnaire every 3 months. Patients with an estimated Glomerular Filtration Rate (eGFR) < 40mL/min are randomized into three groups of follow-up

1. PRO-based follow-up (The clinicians use the PRO data to decide whether a patient needs a visit or not)
2. PRO-based telephone consultations (The clinician use the PRO-data to support the communication with the patient)
3. Usual outpatient follow-up visits (Patients are seen in the outpatient clinic)

The aim of this study is to compare the effect on the clinical outcomes, the utilisation of resources, and patient-reported outcome in three types of follow-up in a non-inferiority randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the renal care services at Aarhus University Hospital or Regional Hospital Central Jutland, Viborg
* Estimated Glomerular Filtration Rate (eGFR) between 10-39 mL/min 1.73m2.
* Aged ≥18 years old
* Ability to provide fully informed written consent for participation in the study

Exclusion Criteria:

* Patients unwilling to participate in PRO-based follow-up
* Patients who, in the opinion of the consenting professional, cannot speak, read or write Danish sufficiently well to complete the PRO questionnaire unaided
* Patients with hearing disabilities
* Patients with an eGFR > 39mL/min 1.73m2 at their first visit at the hospital
* Patients who have received (or have a scheduled date to receive) a kidney transplant
* A terminal illness that, in the opinion of the consultant assessing eligibility, is likely to lead to the death of the patient within 6 months of starting participation in the study
* Patients receiving chemotherapy, with end stage Chronic Obstructive Lung disease, or with heart failure with Ejection Fraction (EF)< 15 %.
* A projected risk of progression to end-stage renal failure within 6 months, determined from albumin/creatinine ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Estimated Glomerular Filtration Rate (eGFR) at 18 months | Measured at baseline, 6, 12 and 18 months after randomisation
  Measurement for renal function

SECONDARY OUTCOMES:
Mortality | 18 months after randomization
  Overall mortality
End Stage Renal Disease (ESRD) | 18 months after randomization
  Has the patient initiated dialyses during follow-up, Hemodialysis, peritoneal dialysis
Kidney transplantation | 18 months after randomization
  Has the patient received a kidney transplant during follow-up
Hospital admission | From baseline at 18 months after randomization
  Difference in number of admissions
Number of contacts | 18 months after randomization
  Number of contacts includes all contacts with the outpatient clinic in the study follow-up period
General Health (SF36), | Baseline, 6,12 and 18 months after randomization
  General health will be assessed by items from the SF-36 questionnaire
Illness perception (BIPQ) | Baseline, 6,12 and 18 months after randomization
  Illness perception will be assessed by the Brief Illness perception questionnaire
Quality of Life (EQ-5D) | Baseline, 6,12 and 18 months after randomization
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention
Satisfaction with care | 6,12,18 months after randomization
  Satisfaction will be assessed by one item from the Danish Cancer Society Patient reported experience measures PREM (Barometer) Questionnaire
Confidence | 6,12,18 months after randomization
  Confidence will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire
Treatment safety | 6,12,18 months after randomization
  Safety will be assessed by one item from the Danish Cancer Society PREM (Barometer) Questionnaire
Patient involvement | Patient involvement will be measured at 6,12 and18 months
  Patient involvement will be assessed by 5 questions from DEFACTUM (Central Denmark Region) Questionnaire

OTHER OUTCOMES:
Baseline questionnaires of non-participants | Baseline questionnaires
  All patients who met the inclusion criteria will be asked to fill in a questionnaire. The questionnaire will include Health Literacy (subscale 4,6,9), Selfefficacy, General Health (SF-36) and 5 renal specific symptoms (KDQOL), Patient activation (2+12), education and employment status. The purpose is to identify baseline differences between participants and non-participants and thereby testing the PRO system for generalizability.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henrik Hjollund, MD,Professor, Study Director — Regional Hospital West Jutland; Birgith Grove, MHSc, Principal Investigator — Aarhus University Hospital & Regional Hospital West Jutland
Locations (1):
- Birgith Engelst Grove, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grove BE, Ivarsen P, de Thurah A, Schougaard LM, Kyte D, Hjollund NH. Remote follow-up using patient-reported outcome measures in patients with chronic kidney disease: the PROKID study - study protocol for a non-inferiority pragmatic randomised controlled trial. BMC Health Serv Res. 2019 Sep 4;19(1):631. doi: 10.1186/s12913-019-4461-y. PMID 31484523
- [Derived] Grove BE, Schougaard LMV, Mose F, Randers E, Hjollund NH, Ivarsen P, De Thurah A. Remote symptom monitoring with patient-reported outcome measures in outpatients with chronic kidney disease (PROKID): a multicentre randomised controlled non-inferiority study. Clin Kidney J. 2024 Jun 14;17(7):sfae176. doi: 10.1093/ckj/sfae176. eCollection 2024 Jul. PMID 39006159
- [Derived] Grove BE, de Thurah A, Ivarsen P, Kvisgaard AK, Hjollund NH, Grytnes R, Schougaard LMV. Remote Symptom Monitoring Using Patient-Reported Outcomes in Patients With Chronic Kidney Disease: Process Evaluation of a Randomized Controlled Trial. JMIR Form Res. 2024 Apr 24;8:e48173. doi: 10.2196/48173. PMID 38656781
- Available data/document: Study Protocol: 31484523 — https://pubmed.ncbi.nlm.nih.gov/31484523/ — Data can be accessed by request from the corresponding author